CLINICAL TRIAL: NCT01585649
Title: Multicenter, Open-label Study to Assess the Pharmacokinetics (PK), Pharmacodynamics (PD), Efficacy, Safety, Tolerability, and Immunogenicity of a Single, Subcutaneous Dose of 100µg/kg XM22 in 21 Children With Ewing Family of Tumors or Rhabdomyosarcoma
Brief Title: PK/PD of XM22 in Children With Ewing Family of Tumors or Rhabdomyosarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merckle GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: XM22-07; 2011-004742-18 (EudraCT Number)
Record Dates: First submitted 2012-04-18; First posted 2012-04-26 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Ewing Family of Tumors, Rhabdomyosarcoma
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral; Rhabdomyosarcoma | interventions — pegfilgrastim

ARMS (1):
- XM22, 100 μg/kg BW (Experimental)
  Interventions: Drug: Lipegfilgrastim

INTERVENTIONS:
Drug: Lipegfilgrastim — Lipegfilgrastim 100ug/kg

SUMMARY:
This is a Phase I, open label study aimed at assessing the pharmacokinetics, pharmacodynamics, the efficacy, safety, and tolerability of a single injection of XM22 in children with Ewing family of tumors or rhabdomyosarcoma scheduled to receive chemotherapy (CTX)

ELIGIBILITY:
Inclusion Criteria:

* Male or female children and adolescents aged 2 to <18 years
* Written informed consent provided by parent(s)/legal representative(s) of the pediatric patient and patient's assent if appropriate
* Able to understand and/or follow study instructions alone or with parental assistance
* Diagnosed with the Ewing family of tumors or Rhabdomyosarcoma
* Scheduled to receive 1 of the following CTX regimens (inpatient or outpatient)
* For the Ewing family of tumors:

  * vincristine/ifosfamide/doxorubicin/etoposide (VIDE); with concomitant sodium 2-mercaptoethane sulfonate (MESNA) according to local standards
  * vincristine/doxorubicin/cyclophosphamide alternating with ifosfamide/etoposide (VDC/IE); with concomitant MESNA treatment according to local standards
* For rhabdomyosarcoma:

  * vincristine/actinomycin/cyclophosphamide (VAC)
  * vincristine/doxorubicin/cyclophosphamide alternating with ifosfamide/etoposide (VDC/IE); with concomitant MESNA treatment according to local standards
* Chemotherapy-naïve
* Body weight ≥15 kg
* White blood cell (WBC) count >2.5 x 109/L, absolute neutrophil count (ANC) ≥1.5 x 109/L, and platelet count ≥100 x 109/L (at screening and prior to CTX)
* For patients aged ≥12 years, Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (See Appendix A.)
* Fertile patients (male or female) must use highly reliable contraceptive measures (i.e. two of the following: oral contraception, implants, injections, barrier contraception, and intrauterine device, or vasectomized/sterilized partners, or sexual abstinence). For purposes of this study, a fertile female patient is any female patient who has experienced menarche and who has not undergone tubal ligation.
* Female patients who have attained menarche must have a negative urine pregnancy test at the screening visit.

Exclusion Criteria:

* Previous exposure to filgrastim, pegfilgrastim or lenograstim or other G-CSFs in clinical development within 6 months prior to the XM22 administration
* Known hypersensitivity to filgrastim, pegfilgrastim or lenograstim or any other G-CSF in clinical development
* History of congenital neutropenia or cyclic neutropenia
* Any illness or condition that in the opinion of the Investigator may affect the safety of the patient or the evaluation of any study endpoint
* Pregnant or nursing women
* Fertile patients who do not agree to use highly reliable contraceptive measures during the entire duration of the study
* Prior bone marrow or stem cell transplant, or prior radiation to ≥25% of bone marrow (e.g. whole pelvic radiation) for any reason, or any therapeutic radiation within the 3 weeks prior to the XM22 dose
* Ongoing active infection or history of infectious disease within 2 weeks prior to the screening visit
* Treatment with lithium at screening or planned during the study.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
PK: Area under the curve, Maximum observed serum concentration (Cmax), Rate constant associated with terminal phase, Mean Residence Time, Time to reach Cmax, and Apparent volume of distribution during terminal phase after non-intravenous administration | 16 months
  A total of 7 PK samples will be obtained at prespecified periods

SECONDARY OUTCOMES:
PD:Absolute Neutrophil Count | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Lammerich, MD, Study Director — Merckle GmbH, Teva Ratiopharm
Locations (18):
- Bulgaria (3):
  - Teva Investigational Site 0103, Plovdiv
  - Teva Investigational Site 0101, Sofia
  - Teva Investigational Site 0102, Varna
- Teva Investigational Site 0201, Prague, Czechia
- Teva Investigational Site 0301, Budapest, Hungary
- Teva Investigational Site 0401, Lublin, Poland
- Russia (7):
  - Teva Investigational Site 0501, Chelyabinsk
  - Teva Investigational Site 0507, Krasnodar
  - Teva Investigational Site 0505, Moscow
  - Teva Investigational Site 0506, Moscow
  - Teva Investigational Site 0508, Moscow
  - Teva Investigational Site 0502, Saint Petersburg
  - Teva Investigational Site 0504, Yekaterinburg
- Ukraine (5):
  - Teva Investigational Site 0701, Dnipropetrovsk
  - Teva Investigational Site 0705, Donetsk
  - Teva Investigational Site 0702, Kharkiv
  - Teva Investigational Site 0704, Kyiv
  - Teva Investigational Site 0703, Lviv